CLINICAL TRIAL: NCT07257744
Title: A Comparative Evaluation of Intravenous Analgesia, Thoracic Epidural Analgesia, and Erector Spinae Plane Block on Chronic Postoperative Pain Following Open Heart Surgery
Brief Title: Comparison of IV Analgesia, Thoracic Epidural Analgesia, and ESP Block for Chronic Pain After Open Heart Surgery
Acronym: TEA-ESPB-IV
Status: Recruiting | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, Associate Professor of Anesthesiology and Reanimation, Karadeniz Technical University
Other Study IDs: KTU-ANES-CHRONICPAIN-2024-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Postoperative Pain; Open Heart Surgery; Postoperative Analgesia; Analgesia
Keywords: Open Heart Surgery; Chronic Postoperative Pain; Post-Sternotomy Pain; Thoracic Epidural Analgesia (TEA); Erector Spinae Plane Block (ESPB); Pain Management; Cardiac Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Analgesia; Tea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intravenous Analgesia Group (IV): Participants who receive routine postoperative intravenous analgesia (opioid and/or non-opioid medications) as determined by the clinical anesthesia team. No protocol-assigned intervention is applied; analgesia is selected based on routine clinical practice.
  Interventions: Other: Intravenous Analgesia; Other: Thoracic Epidural Analgesia (TEA); Other: Erector Spinae Plane Block (ESPB)
- Thoracic Epidural Analgesia Group (TEA): Participants who receive thoracic epidural analgesia via an epidural catheter placed preoperatively for postoperative pain control. TEA is administered according to institutional routine practice and is not assigned by the study protocol
  Interventions: Other: Intravenous Analgesia; Other: Thoracic Epidural Analgesia (TEA); Other: Erector Spinae Plane Block (ESPB)
- Erector Spinae Plane Block Group (ESPB): Participants who receive bilateral erector spinae plane block (ESPB) performed preoperatively for postoperative analgesia. This block is a routine clinical procedure and is not assigned or modified by the study protocol.
  Interventions: Other: Intravenous Analgesia; Other: Thoracic Epidural Analgesia (TEA); Other: Erector Spinae Plane Block (ESPB)

INTERVENTIONS:
Other: Intravenous Analgesia — Routine postoperative intravenous analgesia (opioid and/or non-opioid medications) administered according to standard clinical care. This is not assigned by protocol and represents usual practice.
  Other Names: IV Analgesia; Intravenous Pain Management
Other: Thoracic Epidural Analgesia (TEA) — Thoracic epidural catheterization performed as part of routine postoperative analgesia management. This practice is determined by the clinical anesthesia team and not assigned by the study protocol.
Other: Erector Spinae Plane Block (ESPB) — Bilateral erector spinae plane block performed preoperatively as part of routine perioperative analgesia. The technique is applied at the discretion of the clinical anesthesia team and is not protocol-assigned.

SUMMARY:
This prospective observational study aims to compare three routinely used postoperative analgesia techniques in patients undergoing open heart surgery: intravenous analgesia, thoracic epidural analgesia (TEA), and bilateral erector spinae plane block (ESPB). The primary objective is to evaluate the impact of these analgesia modalities on the development of chronic postoperative pain at 3 months. Secondary objectives include assessing postoperative acute pain scores, additional analgesic requirements, extubation time, mobilization time, intensive care unit stay, hospital stay, respiratory complications, and the relationship between acute and chronic pain. No intervention is assigned by protocol, and all analgesia methods are applied as part of routine clinical practice.

DETAILED DESCRIPTION:
This prospective observational study is designed to evaluate and compare three commonly used postoperative analgesia modalities in adult patients undergoing open heart surgery through median sternotomy: intravenous analgesia, thoracic epidural analgesia (TEA), and bilateral erector spinae plane block (ESPB). All analgesia techniques included in this study represent routine clinical practices performed by the anesthesia team, and no intervention is assigned according to a research protocol. Patients receive whichever analgesia method is chosen by the clinical anesthesia team based on individual clinical conditions. Thus, the study reflects real-world practice in a single tertiary cardiac surgery center.

The primary objective is to determine the effect of these analgesia methods on the development of chronic postoperative pain at 3 months following surgery. Chronic pain will be assessed using the Numeric Rating Scale (NRS) and the S-LANSS questionnaire, administered either via telephone or in-person follow-up. Secondary objectives include the evaluation of postoperative acute pain scores, additional analgesic consumption, extubation time, mobilization time, intensive care unit (ICU) length of stay, hospital length of stay, respiratory parameters, complications such as reintubation or need for non-invasive mechanical ventilation, bronchodilator use, sedation requirements, urine output, and perioperative hemodynamic stability. The study also aims to analyze the correlation between acute postoperative pain and subsequent chronic pain development.

Eligible patients are those aged 18-85 years, classified as ASA I-III, with a body mass index (BMI) below 35 kg/m², and scheduled for open heart surgery at Karadeniz Technical University Farabi Hospital. Exclusion criteria include coagulation disorders, infection at the intervention site, psychiatric disorders, chronic pain treatment, allergy to anesthetic agents, inability to cooperate or communicate, prior open heart surgery, chronic analgesic or antidepressant use, and significant comorbid conditions affecting participation.

Patients included in the study will have their perioperative data extracted from anesthesia records, ICU follow-up forms, and hospital medical charts. Routine postoperative pain measurements will be performed using the NRS. No additional procedures, medications, or interventions beyond routine care will be conducted.

The study aims to enroll 90 patients (30 per group). Data will be analyzed using Statistical Package for the Social Sciences (SPSS). Normality will be assessed using the Kolmogorov-Smirnov test. Parametric and nonparametric tests, including Student's t-test, Mann-Whitney U, chi-square test, repeated-measures ANOVA, and Friedman test, will be used as appropriate. A significance level of p < 0.05 will be accepted.

This study is expected to contribute to the understanding of analgesic strategies in cardiac surgery and their role in preventing chronic postoperative pain, improving recovery, and reducing complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 85 years
* Classified as ASA physical status I-III
* Scheduled to undergo open heart surgery with median sternotomy
* BMI < 35 kg/m²
* Able to understand and provide written informed consent
* Eligible to receive any of the routine analgesia methods (intravenous analgesia, thoracic epidural analgesia, or erector spinae plane block)

Exclusion Criteria:

* Age < 18 or > 85 years
* BMI ≥ 35 kg/m²
* Coagulation disorders
* Infection at the intervention site
* Known allergy to local anesthetics or induction agents
* Psychiatric disorders limiting cooperation
* Use of chronic pain medications, antidepressants, corticosteroids, antiepileptics, or routine analgesics
* Inability to cooperate, communicate, or follow commands
* Physical or verbal performance impairment
* Previous open heart surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 85 years who are scheduled to undergo open heart surgery with median sternotomy at Karadeniz Technical University Farabi Hospital. All participants will receive one of the routinely used postoperative analgesia methods (intravenous analgesia, thoracic epidural analgesia, or erector spinae plane block) as determined by the clinical anesthesia team. Only patients classified as ASA physical status I-III and able to provide informed consent are included. Individuals with major comorbidities that interfere with participation, prior cardiac surgery, chronic pain treatment, or contraindications to routine analgesia methods are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Chronic Postoperative Pain at 3 Months | 3 Months Postoperative
  Chronic postoperative pain will be assessed 3 months after surgery using the Numeric Rating Scale (NRS, 0-10) and the S-LANSS questionnaire. Participants will be contacted via telephone or in-person follow-up. Chronic pain is defined as pain persisting beyond the expected healing period and lasting at least 3 months.

SECONDARY OUTCOMES:
Acute Postoperative Pain Scores | 0-72 hours postoperative
  Pain intensity will be measured using the Numeric Rating Scale (NRS, 0-10) at routine postoperative intervals in the ICU and ward.
Additional Analgesic Consumption | 0-72 hours postoperative
  Total amount and frequency of rescue analgesic medications administered during the postoperative hospital period.
Extubation Time | Up to 72 hours postoperative
  Time from ICU admission after surgery to successful extubation, recorded from anesthesia and ICU charts.
Mobilization Time | Postoperative day 0-2
  Time to first mobilization (sitting, standing, or ambulation) recorded by ICU or ward nursing staff.
ICU Length of Stay | Up to 7 days
  Duration of ICU stay in hours, extracted from patient records.
Hospital Length of Stay | Up to 14 days
  Total hospitalization duration from surgery to discharge.
Postoperative Respiratory Events | Up to 14 days postoperative
  Incidence of re-intubation, need for non-invasive mechanical ventilation (NIMV), bronchodilator therapy, or respiratory complications.
Correlation Between Acute and Chronic Pain | From immediate postoperative period to 3-month follow-up
  Correlation analysis between early postoperative pain scores (NRS) and chronic pain severity (NRS + S-LANSS) at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Farabi Hospital, Trabzon, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study is based on clinical follow-up data collected for a single-center observational thesis project, and no data sharing plan has been established.

REFERENCES:
- [Background] Yu H, Zheng JQ, Hua YS, Ren SF, Yu H. Influence of volatile anesthesia versus total intravenous anesthesia on chronic postsurgical pain after cardiac surgery using the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials criteria: study protocol for a prospective randomized controlled trial. Trials. 2019 Nov 27;20(1):645. doi: 10.1186/s13063-019-3742-4. PMID 31775854
- [Background] Martorella G, McDougall GJ Jr. Barriers and Facilitators to the Prevention of Chronic Pain in the Subacute Phase After Cardiac Surgery. Pain Manag Nurs. 2021 Feb;22(1):28-35. doi: 10.1016/j.pmn.2020.09.004. Epub 2020 Nov 11. PMID 33189543
- [Background] Yan H, Chen W, Chen Y, Gao H, Fan Y, Feng M, Wang X, Tang H, Yin J, Qian Y, Ding M, Cang J, Miao C, Wang H. Opioid-Free Versus Opioid-Based Anesthesia on Postoperative Pain After Thoracoscopic Surgery: The Use of Intravenous and Epidural Esketamine. Anesth Analg. 2023 Aug 1;137(2):399-408. doi: 10.1213/ANE.0000000000006547. Epub 2023 Jul 14. PMID 37267129
- [Background] Elsharkawy H, Clark JD, El-Boghdadly K. Evidence for regional anesthesia in preventing chronic postsurgical pain. Reg Anesth Pain Med. 2025 Feb 5;50(2):153-159. doi: 10.1136/rapm-2024-105611. PMID 39909548